CLINICAL TRIAL: NCT03449251
Title: A Series of Pilot Studies to Evaluate the Haemodynamic and Metabolic Effects of Apelin and Relaxin in Healthy Humans, Subjects With Increased Weight and Patients With Type 2 Diabetes Mellitus
Brief Title: A Series of Pilot Studies to Evaluate the haemoDynamic and mEtabolic Effects oF apelIn aNd rElaxin
Acronym: DEFINE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); AstraZeneca (Industry); MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Joseph Cheriyan, MD, Consultant Physician & Clinical Pharmacologist/Assoc Lecturer, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: DEFINE (A094666)
Record Dates: First submitted 2018-02-06; First posted 2018-02-28 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes Mellitus
Keywords: Apelin; Relaxin
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2 | interventions — Apelin; Relaxin; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Identical, colourless solution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Substudy 1A - Apelin (Experimental): In sub-study 1A Healthy participants will receive systemic infusions of Apelin to establish a dose range
  Interventions: Drug: Apelin
- Substudy 1B - Apelin/Normal Saline (Experimental): In sub-study 1B , individuals with Type 2 Diabetes and individuals with increase weight will receive systemic infusions of Apelin or Normal Saline
  Interventions: Drug: Apelin; Drug: Normal saline
- Substudy 2A - Relaxin/Normal Saline (Experimental): In sub-study 2A Healthy participants will receive intra-arterial infusions of Relaxin
  Interventions: Drug: Relaxin; Drug: Normal saline
- Substudy 2B - Relaxin (Experimental): In sub-study 2B Healthy participants will receive intra-arterial infusions of Relaxin followed by verapamil (on a background infusion of either LN Monomethyl Arginine or Normal Saline, to test effects on nitric oxide)
  Interventions: Drug: Relaxin; Diagnostic Test: Verapamil; Diagnostic Test: LN Monomethyl arginine
- Substudy 3A - Relaxin with Apelin/Saline (Experimental): In sub-study 3A Healthy participants will receive intra-arterial infusions of Relaxin (background infusion apelin/Normal Saline)
  Interventions: Drug: Apelin; Drug: Relaxin; Drug: Normal saline
- Substudy 3B - Apelin with Relaxin/Saline (Experimental): In sub-study 3B Healthy participants will receive intra-arterial infusions of Apelin (background infusion Relaxin/Normal Saline)
  Interventions: Drug: Apelin; Drug: Relaxin; Drug: Normal saline
- Substudy 4 - Apelin and Relaxin (Experimental): In sub-study 4 Healthy participants, Individuals with Type 2 Diabetes and Individuals with increase weight will receive systemic infusions of Normal saline, Relaxin, Apelin and relaxin
  Interventions: Drug: Apelin; Drug: Relaxin
- Substudy 5 - Relaxin/Saline (Experimental): In sub-study 5 Healthy participants will be allocated to 1 of 4 Relaxin dosing groups and will receive dorsal hand vein infusion of 3 incremental doses of Normal Saline/ D5W and Relaxin
  Interventions: Drug: Relaxin; Drug: Normal saline

INTERVENTIONS:
Drug: Apelin — Apelin is an endogenous peptide that activate a single G-protein couple receptor. Apelin inhibits insulin secretion, decreases glucose levels and increases insulin sensitivity.
  Arms: Substudy 1A - Apelin; Substudy 1B - Apelin/Normal Saline; Substudy 3A - Relaxin with Apelin/Saline; Substudy 3B - Apelin with Relaxin/Saline; Substudy 4 - Apelin and Relaxin
Drug: Relaxin — Relaxin is RLN2 encoded endogenous peptide hormone, which binds to G protein coupled receptor RXFP1.
  Other Names: RLX
  Arms: Substudy 2A - Relaxin/Normal Saline; Substudy 2B - Relaxin; Substudy 3A - Relaxin with Apelin/Saline; Substudy 3B - Apelin with Relaxin/Saline; Substudy 4 - Apelin and Relaxin; Substudy 5 - Relaxin/Saline
Drug: Normal saline — Vehicle
  Other Names: Saline
  Arms: Substudy 1B - Apelin/Normal Saline; Substudy 2A - Relaxin/Normal Saline; Substudy 3A - Relaxin with Apelin/Saline; Substudy 3B - Apelin with Relaxin/Saline; Substudy 5 - Relaxin/Saline
Diagnostic Test: Verapamil — NO independent challenge agent
  Arms: Substudy 2B - Relaxin
Diagnostic Test: LN Monomethyl arginine — Basal NO synthase inhibitor
  Other Names: LNMMA
  Arms: Substudy 2B - Relaxin

SUMMARY:
Type two diabetes mellitus (T2DM) is a common, long term metabolic disorder characterised by hyperglycaemia (high blood glucose) resulting from insulin resistance and relative insulin insufficiency. The risk of developing insulin resistance and subsequently T2DM is increased by being overweight and also through a sedentary lifestyle. As the onset can be gradual, physiological damage may have occurred prior to diagnosis. Diabetes is associated with the development of microvascular complications (diabetic nephropathy, neuropathy, and retinopathy), and macrovascular complications (coronary artery disease, peripheral arterial disease, and stroke). While there are many treatments available for T2DM, these complications may still arise, leading to significant morbidity and mortality. There is therefore an urgent need to identify novel signalling pathways that may contribute to the development of diabetes related complications. The identification of these pathways may ultimately lead to the development of new therapies targeting better blood glucose control and preventing these subsequent complications.

Both animal and human studies have indicated that two endogenous peptides, apelin and relaxin both act as vasodilators in the human cardiovascular system and could also have beneficial action in T2DM. Therefore, we aim to carry out experimental medicine studies to test this hypothesis, and explore the signalling pathway in the human vascular system.

DETAILED DESCRIPTION:
An extensive body of evidence demonstrates a direct association between T2DM and cardiovascular complications and mortality. Unfortunately, current therapies for diabetes have failed to be translated into improvements in cardiovascular outcomes, highlighting an urgent need to develop novel therapeutic strategies that can ultimately achieve the dual outcome of improving glycaemic control and improving cardiovascular function.

While the precise cellular mechanisms involved remain to be elucidated, we hypothesise that the apelin and relaxin pathways meet these two criteria and therefore are potential therapeutic targets in conditions of abnormal glucose metabolism and heart failure.

Apelin and relaxin are safe for parenteral use as they are naturally occurring peptide hormones, have a short half-life and will be rapidly cleared. They target endogenous receptors and post-receptor signalling, and have been used in human trials without any significant side effects reported.

ELIGIBILITY:
Inclusion Criteria:

Healthy participants

* Have given written informed consent to participate
* Aged 18 to 70 years inclusive
* Male or female
* Current non-smoker
* If female, either postmenopausal or on days 2-9 of menstrual cycle and negative pregnancy test performed on the day of the of visit
* BMI in range for studies 1 and 4: 18.5-24.9 kg/m2 with waist circumference lower than 88 centimetres (35 inches) for women or 102 cm (40 inches) for men, and/or body fat level less than 32 % for women or 25% for men
* BMI in range for studies 2 and 3: 18.5-30.0 kg/m2 without limitations in waist circumference or body fat level

Overweight/obese participants

* Have given written informed consent to participate
* Aged 18 to 70 years inclusive
* Male or female
* Current non-smoker
* If female, either postmenopausal or on days 2-9 of menstrual cycle and negative pregnancy test performed on the day of the of visit
* BMI in range of 25-34.9 kg/m2 (inclusive) with either waist circumference higher than 88cm (35 inches) for women or 102 cm (40 inches) for men, and/or body fat levels in excess of 32% for women or 25% for men

Participants with type 2 diabetes mellitus

* Have given written informed consent to participate
* Aged 18 to 70 years inclusive
* Male or female
* Current non-smoker
* If female, either postmenopausal or on days 2-9 of menstrual cycle and negative pregnancy test performed on the day of the of visit
* BMI in range of 25-34.9 kg/m2 (inclusive) with either waist circumference higher than 88cm (35 inches) for women or 102 cm (40 inches) for men, and/or body fat levels in excess of 32% for women or 25% for men
* Documented diagnosis of Type 2 Diabetes Mellitus, either diet controlled or treated with oral hypoglycaemic therapy

Exclusion Criteria:

* Hypersensitivity to any of the study drugs or excipients
* Systemic Hypertension (sustained BP >160/100mmHg) or hypotension (systolic BP below 90 mmHg)
* Known heart disease
* Implanted heart pace-maker or implantable cardioverter defibrillator (ICD)
* Known active malignancy
* Known renal failure (creatinine >140µmol/L)
* Known neurological disease
* History of Scleroderma (Study 4 only)
* Current pregnancy, breast feeding
* Use of vasoactive medications or NSAIDS/aspirin within 24 hours of study visits
* Use of caffeine within 24 hours of study visits
* Current involvement in the active treatment phase of other research studies, (excluding observations/non-interventional)
* Second or third-degree AV block, sino-atrial block, sick sinus syndrome or sinus bradycardia
* Known HIV, hepatitis B or C
* Needle phobia
* Participants treated with formal anticoagulant therapy such as, but not limited to, heparin, warfarin or clopidogrel
* Diagnosis of Type 1 Diabetes Mellitus or current usage of insulin or other injectable drugs for the treatment of diabetes such as but not limited to GLP1 agonists
* BMI <18.5
* Aged <18 or >70 years
* Any other clinical reason which may preclude entry in the opinion of the investigator

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Sub-study 1a: Changes in markers of glucose homeostasis in healthy participants after infusion of apelin (Glucose) | Visit 2 to visit 4, over a period of up to 8 weeks
  Glucose, in mmol/l
Sub-study 1a: Changes in markers of glucose homeostasis in healthy participants after infusion of apelin (C-Peptide) | Visit 2 to visit 4, over a period of up to 8 weeks
  C-peptide, in pmol/L
Sub-study 1a: Changes in markers of glucose homeostasis in healthy participants after infusion of apelin (Glucagon) | Visit 2 to visit 4, over a period of up to 8 weeks
  Glucagon, in pg/ml
Sub-study 1a: Changes in markers of glucose homeostasis in healthy participants after infusion of apelin (Insulin) | Visit 2 to visit 4, over a period of up to 8 weeks
  Insulin, in pmol/L
Sub-study 1a: Changes in markers of glucose homeostasis in healthy participants after infusion of apelin (TNF-alpha) | Visit 2 to visit 4, over a period of up to 8 weeks
  TNF-alpha, in pg/ml
Sub-study 1b: Changes in markers of glucose homeostasis in participants with increased weight and participants with type 2 diabetes mellitus after infusion of apelin with or without mixed meal tolerance in obese/overweight and T2DM participants | Visit 2 to visit 5, over a period of up to 14 weeks
  Glucose, in mmol/l
Sub-study 1b: Changes in markers of glucose homeostasis in participants with increased weight and participants with type 2 diabetes mellitus after infusion of apelin with or without mixed meal tolerance in obese/overweight and T2DM participants | Visit 2 to visit 5, over a period of up to 14 weeks
  C-peptide, in pmol/L
Sub-study 1b: Changes in markers of glucose homeostasis in participants with increased weight and participants with type 2 diabetes mellitus after infusion of apelin with or without mixed meal tolerance in obese/overweight and T2DM participants | Visit 2 to visit 5, over a period of up to 14 weeks
  Glucagon, in pg/ml
Sub-study 1b: Changes in markers of glucose homeostasis in participants with increased weight and participants with type 2 diabetes mellitus after infusion of apelin with or without mixed meal tolerance in obese/overweight and T2DM participants | Visit 2 to visit 5, over a period of up to 14 weeks
  Insulin, in pmol/L
Sub-study 1b: Changes in markers of glucose homeostasis in participants with increased weight and participants with type 2 diabetes mellitus after infusion of apelin with or without mixed meal tolerance in obese/overweight and T2DM participants | Visit 2 to visit 5, over a period of up to 14 weeks
  TNF-alpha, in pg/ml
Sub-study 2a: Change in forearm blood flow parameters in healthy participants after infusion of relaxin (Absolute Flow) | Within visit 2, over a period of up to 4 weeks
  Absolute flow in the infused arm, in mg/dL/min
Sub-study 2a: Change in forearm blood flow parameters in healthy participants after infusion of relaxin (Percentage Change) | Within visit 2, over a period of up to 4 weeks
  Percentage change in the infused arm, in %
Sub-study 2a: Change in forearm blood flow parameters in healthy participants after infusion of relaxin (Ratio) | Within visit 2, over a period of up to 4 weeks
  Ratio, expressed as a number (no units as this is a ratio)
Sub-study 2b: Change in forearm blood flow parameters in healthy participants after infusion of relaxin in the presence of L-NMMA or normal saline | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio; absolute flow and percentage change in the infused arm
Sub-study 2b: Change in forearm blood flow parameters in health participants after infusion of verapamil in the presence of L-NMMA or normal saline (Ratio) | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio; expressed as a number (no units as this is a ratio)
Sub-study 2b: Change in forearm blood flow parameters in health participants after infusion of verapamil in the presence of L-NMMA or normal saline (Absolute Flow) | Visit 2 to visit 3, over a period of up to 10 weeks
  Absolute flow in the infused arm, in mg/dL/min
Sub-study 2b: Change in forearm blood flow parameters in health participants after infusion of verapamil in the presence of L-NMMA or normal saline (Percentage Change) | Visit 2 to visit 3, over a period of up to 10 weeks
  Percentage change in the infused arm, In %
Sub-Study 3a: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial relaxin in the presence of apelin | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio; absolute flow and percentage change in the infused arm
Sub-Study 3a: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial relaxin in the presence of apelin (Ratio) | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio, expressed as a number (no units as this is a ratio)
Sub-Study 3a: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial relaxin in the presence of apelin (Absolute Flow) | Visit 2 to visit 3, over a period of up to 10 weeks
  Absolute flow in the infused arm, in mg/dL/min
Sub-Study 3a: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial relaxin in the presence of apelin (Percentage Change) | Visit 2 to visit 3, over a period of up to 10 weeks
  Percentage change in the infused arm, In %
Sub-Study 3b: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial apelin in the presence of relaxin (Ratio) | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio, expressed as a number (no units as this is a ratio)
Sub-Study 3b: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial apelin in the presence of relaxin (Absolute Flow) | Visit 2 to visit 3, over a period of up to 10 weeks
  Absolute flow in the infused arm, in mg/dL/min
Sub-Study 3b: Change in forearm blood flow parameters in healthy participants after incremental infusions of intra-arterial apelin in the presence of relaxin (Percentage Change) | Visit 2 to visit 3, over a period of up to 10 weeks
  Percentage change in the infused arm, In %
Sub-study 4: Changes in markers of glucose homeostasis healthy participants, participants with increased weight and participants with type 2 diabetes mellitus after infusion of relaxin with and without apelin (Glucose) | Visit 2 to Visit 4, over a period of up to 8 weeks
  Glucose, in each of the groups, in mmol/L
Sub-study 4: Changes in markers of glucose homeostasis healthy participants, participants with increased weight and participants with type 2 diabetes mellitus after infusion of relaxin with and without apelin (C-peptide) | Visit 2 to Visit 4, over a period of up to 8 weeks
  C-peptide, in each of the groups, in pmol/L
Sub-study 4: Changes in markers of glucose homeostasis healthy participants, participants with increased weight and participants with type 2 diabetes mellitus after infusion of relaxin with and without apelin (Glucagon) | Visit 2 to Visit 4, over a period of up to 8 weeks
  glucagon, in each of the groups,in pg/ml
Sub-study 4: Changes in markers of glucose homeostasis healthy participants, participants with increased weight and participants with type 2 diabetes mellitus after infusion of relaxin with and without apelin (Insulin) | Visit 2 to Visit 4, over a period of up to 8 weeks
  Insulin, in each of the groups, in pmol/L
Sub-study 4: Changes in markers of glucose homeostasis healthy participants, participants with increased weight and participants with type 2 diabetes mellitus after infusion of relaxin with and without apelin (TNF-alpha) | Visit 2 to Visit 4, over a period of up to 8 weeks
  TNF-alpha, in each of the groups, in pg/ml
Sub-study 5: Change in hand vein diameter after relaxin infusion in healthy participants | Visit 2
  Hand vein Demeter is measured using Aellig dorsal hand vein technique

SECONDARY OUTCOMES:
Sub-study 1a: Changes in parameters of cardiovascular haemodynamics in healthy participants after infusion of apelin (Echocardiography) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Echocardiography, in L/min
Sub-study 1a: Changes in parameters of cardiovascular haemodynamics in healthy participants after infusion of apelin (Innocor) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Innocor, in L/min
Sub-study 1a: Changes in parameters of cardiovascular haemodynamics in healthy participants after infusion of apelin (Bioimpedance) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by bioimpedance, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin (Echocardiography) | VIsit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Echocardiography, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin (Innocor) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Innocor, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin (Bioimpedance) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by bioimpedance, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin,after a mixed meal challenge (Echocardiography) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Echocardiography, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin, after a mixed meal challenge (Innocor) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Innocor, in L/min
Sub-study 1b: Changes in parameters of cardiovascular haemodynamics in obese/overweight and T2DM participants after infusion of apelin,after a mixed meal challenge (Bioimpedance) | VIsit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by bioimpedance, in L/min
Sub-study 1b: Changes in markers of glucose homeostasis after infusion of apelin in obese/overweight and T2DM, after a mixed meal challenge (Clugose) | Visit 2 to visit 5, over a period of up to 14 weeks
  Glucose, in mmol/L
Sub-study 1b: Changes in markers of glucose homeostasis after infusion of apelin in obese/overweight and T2DM, after a mixed meal challenge (C-peptide) | Visit 2 to visit 5, over a period of up to 14 weeks
  C-peptide, in pmol/L
Sub-study 1b: Changes in markers of glucose homeostasis after infusion of apelin in obese/overweight and T2DM, after a mixed meal challenge (Glucagon) | Visit 2 to visit 5, over a period of up to 14 weeks
  Glucagon, in pg/ml
Sub-study 1b: Changes in markers of glucose homeostasis after infusion of apelin in obese/overweight and T2DM, after a mixed meal challenge (Insulin) | Visit 2 to visit 5, over a period of up to 14 weeks
  Insulin, in pmol/L
Sub-study 1b: Changes in markers of glucose homeostasis after infusion of apelin in obese/overweight and T2DM, after a mixed meal challenge (TNF alpha) | Visit 2 to visit 5, over a period of up to 14 weeks
  TNF alpha, in pg/ml
Sub-study 2b: Change in forearm blood flow parameters after infusion of verapamil in the presence of L-NMMA or saline (Ratio) | Visit 2 to visit 3, over a period of up to 10 weeks
  Ratio,expressed as a number (no units as this is a ratio)
Sub-study 2b: Change in forearm blood flow parameters after infusion of verapamil in the presence of L-NMMA or saline (Absolute Flow) | Visit 2 to visit 3, over a period of up to 10 weeks
  Absolute flow in the infused arm, in mg/dL/min
Sub-study 2b: Change in forearm blood flow parameters after infusion of verapamil in the presence of L-NMMA or saline (Percentage Change) | Visit 2 to visit 3, over a period of up to 10 weeks
  Percentage change in the infused arm, In %
Sub-study 4: Change in cardiovascular haemodynamics after infusion of relaxin (Echocardiography) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Echocardiography, in L/min
Sub-study 4: Change in cardiovascular haemodynamics after infusion of relaxin (Bioimpedance) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by bioimpedance, in L/min
Sub-study 4: Change in cardiovascular haemodynamics after infusion of relaxin (Innocor) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Innocor, in L/min
Sub-study 4: Change in cardiovascular haemodynamics after combined infusion of relaxin and apelin (Echocardiography) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Echocardiography, in L/min
Sub-study 4: Change in cardiovascular haemodynamics after combined infusion of relaxin and apelin (Bioimpedance) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by bioimpedance, in L/min
Sub-study 4: Change in cardiovascular haemodynamics after combined infusion of relaxin and apelin (Innocor) | Visit 2 to visit 4, over a period of up to 8 weeks
  Cardiac output measured by Innocor, in L/min
Sub-study 4: Change in glucose homeostasis after combined infusion of relaxin and apelin (Glucose) | Visit 2 to visit 4, over a period of up to 8 weeks
  Glucose, in mmol/L
Substudy 4: Change in glucose homeostasis after combined infusion of relaxin and apelin (C-peptide) | Visit 2 to visit 4, over a period of up to 8 weeks
  C-peptide, in pmol/L
Sub-study 4: Change in glucose homeostasis after combined infusion of relaxin and apelin (Glucagon) | Visit 2 to visit 4, over a period of up to 8 weeks
  Glucagon, in pg/ml
Sub-study 4: Change in glucose homeostasis after combined infusion of relaxin and apelin (Insulin) | Visit 2 to visit 4, over a period of up to 8 weeks
  Insulin, in pmol/L
Sub-study 4: Change in glucose homeostasis after combined infusion of relaxin and apelin (TNF alpha) | Visit 2 to visit 4, over a period of up to 8 weeks
  TNF alpha, glucose homeostasis

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBCHB, FRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided